CLINICAL TRIAL: NCT00001544
Title: Genetic Aspects of Neurologic and Psychiatric Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960060; 96-M-0060
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Bipolar Disorder; Mental Disorder Diagnosed in Childhood; Mental Retardation; Schizophrenia
Keywords: DNA Probes; Trinucleotide Repeats; Family Studies; Lymphoblast Cell Lines; Genotyping; Bipolar Affective Disorders; Schizophrenia; Mental Retardation; Neuropsychiatric Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Bipolar Disorder; Intellectual Disability; Schizophrenia

SUMMARY:
The purpose of this study is to improve the understanding of the genetic causes of specific neurologic and psychiatric disorders. The study will focus on conditions of mental retardation, childhood onset schizophrenia, attention deficit hyperactivity disorder (ADHD), atypical psychosis of childhood, and bipolar affective disorder.

The study addresses the belief that there may be several genes contributing to the illness. Researchers intend to use several molecular genetic techniques in order to identify the areas of chromosomes containing genes responsible for the development of these disorders.

Patients will be selected to participate in this study based on an early age of onset of their condition as well as the severity of the illness and the frequency of the illness among family members. Researchers will collect DNA samples from patients as well as affected and unaffected family members of each patient. The DNA samples collected will be analyzed for a variety of genetic abnormalities including; triplet repeat expansions, chromosome rearrangements, and polymorphisms.

DETAILED DESCRIPTION:
We propose to use DNA probes to study patients having specific neurologic and psychiatric disorders, especially focusing on patients with early onset or extreme phenotypes such as childhood onset schizophrenia (COS), mental retardation (MR), attention deficit hyperactivity disorder (ADHD), atypical psychosis of childhood, (multi-dimensional impairment MDI), and bipolar affective disorder (BPAD). This study addresses the hypothesis that genetic risk factors contribute to these diverse phenotypes. Several complementary molecular genetic techniques are employed to identify chromosomal regions containing genes contributing to specific neurologic and psychiatric disorders. Patients will be selected for this study on the basis of the age of onset and severity of neurologic or psychiatric symptoms, familial genetic loading and family structure. Individuals participating in this protocol will be clinically evaluated through other NIMH or NIH clinical protocols, particularly through those of the Child Psychiatry Branch (reference protocol numbers 85-M-0115, 84-M-0050, 97-M-0126). Those subjects meeting inclusion criteria may undergo a screening that may include physical, neurologic or psychiatric examinations. As appropriate, this initial screen may be followed by more formal, structured instruments such as the Schedule for Affective Disorders (SADS), the revised Weschler Adult Intelligence Scale (WAIS-R), the Conner's revised parent and teacher ratings, and the Diagnostic Interview for Children and Adolescents (DICA- version IV) to confirm the clinical diagnosis at the discretion of the treating physician. Venipuncture and/or buccal swabs will be performed in order to obtain samples for DNA extraction or to establish a lymphoblast cell line to be used in genetic tests. Samples will also be collected from family members and controls for these studies.

ELIGIBILITY:
INCLUSION CRITERIA:

Individuals with selected psychiatric and neurologic disorders, including childhood onset schizophrenia, atypical psychosis, mental retardation, bipolar affective disorder, and ADHD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1227
Dates: Start 1996-04; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Willems PJ. Dynamic mutations hit double figures. Nat Genet. 1994 Nov;8(3):213-5. doi: 10.1038/ng1194-213. No abstract available. PMID 7874160
- [Background] Koide R, Ikeuchi T, Onodera O, Tanaka H, Igarashi S, Endo K, Takahashi H, Kondo R, Ishikawa A, Hayashi T, et al. Unstable expansion of CAG repeat in hereditary dentatorubral-pallidoluysian atrophy (DRPLA). Nat Genet. 1994 Jan;6(1):9-13. doi: 10.1038/ng0194-9. PMID 8136840
- [Background] Philibert RA, Hawkins GA, Damschroder-Williams P, Stubblefield BK, Martin BM, Ginns EI. Direct sequencing of trinucleotide repeats from cosmid genomic DNA template. Anal Biochem. 1995 Mar 1;225(2):372-4. doi: 10.1006/abio.1995.1174. No abstract available. PMID 7762809